CLINICAL TRIAL: NCT02722694
Title: A Phase III, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Abatacept 125mg Administered Subcutaneously in Chinese Subjects With Active Rheumatoid Arthritis, Receiving Background Methotrexate, and Experiencing an Inadequate Response to Methotrexate
Brief Title: A Phase 3 Study of Abatacept in Chinese Patients With Active Rheumatoid Arthritis and Inadequate Response to Methotrexate
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-126-III
Record Dates: First submitted 2016-03-10; First posted 2016-03-30 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous(SC) Abatacept (Experimental)
  Interventions: Drug: Subcutaneous(SC) Abatacept; Drug: Methotrexate
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: Subcutaneous(SC) Abatacept — Subjects received 125mg weekly SC abatacept injections for 24 weeks. All subjects who complete 24 weeks double-blind treatment are eligible to enter open label period. During this period, subjects in placebo group will be switched to receive abatacept 125mg administered SC weekly till week 52. Subjects in abatacept group will continue to receive abatacept 125mg weekly.
  Other Names: Orencia
  Arms: Subcutaneous(SC) Abatacept
Other: Placebo — Subjects received weekly SC placebo injections for 24 weeks
  Arms: Placebo
Drug: Methotrexate — All Subjects received backup Methotrexate treatment.

SUMMARY:
The primary objective of this study is to demonstrate superior efficacy of abatacept 125mg administrated SC weekly comparing to placebo after 24 weeks treatment in Chinese subjects who have active rheumatoid arthritis, are receiving methotrexate and experiencing an inadequate response to methotrexate. This will be estimated by the proportion of subjects meeting the American College of Rheumatology (ACR) criteria for 20% improvement (ACR20).

ELIGIBILITY:
Inclusion Criteria:

* Subjects are willing to participate in this study and sign informed consent;
* Subjects must meet the criteria of the America Rheumatism Association (1987) for the diagnosis of rheumatoid arthritis and ACR (1991) functional classes I, II or III;
* Subjects must have had Rheumatoid Arthritis for at least 6 months;
* Subjects who have inadequately response to MTX, must have been taking methotrexate for at least 3 months with minimal dose of 10 mg weekly, and at a stable dose for at least 28 days prior to randomization (Day 1). Methotrexate weekly dose as low as 7.5 mg is permitted for subjects who cannot tolerate higher dose, and the intolerance of higher dose than 7.5mg weekly should be well documented;
* Subjects must have the following disease activity at randomization:

  1. 6 or more swollen joints(66 joint count);
  2. 8 or more tender joints(68 joint count); and
  3. C reactive protein (hsCRP) > 3 mg/L (based on the result of screening visit) or ESR ≥ 28mm/hr;
* All DMARDs (except methotrexate) should be discontinued for at least 28 days prior to study randomization (Day 1), Leflunomide must have been discontinued ≥8 weeks (the subject can be washed-out with cholestyramine according to label recommendations);
* Oral corticosteroid treatment must have been reduced to the prednisone ≤ 10 mg daily or equivalent for 28 days，and stabilized for at least 25 out of 28 days prior to randomization (Day 1). Corticosteroid administered by intra-articular (IA) or intramuscular (IM) will not be allowed 28 days prior to randomization (Day 1);
* Stable NSAIDs are permitted;
* Male and female subject ≥18 years old;
* Women of childbearing potential (WOCBP) must have a negative pregnancy test within 24 hours prior to the start of study medication;

Exclusion Criteria:

* WOCBP and male patients of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 10 weeks after the last dose of study medication;
* Women who are pregnant or breast-feeding;
* Women with a positive pregnancy test on enrollment or prior to study drug administration;
* Subjects meet diagnosis criteria of other rheumatoid disease (e.g., systemic lupus erythematosus);
* Subjects with active vasculitis of the major organ systems (except for subcutaneous rheumatoid nodules);
* Current symptoms of severe, progressive or uncontrolled diseases of renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, neurological, or cerebral. Concomitant medical conditions that, in the opinion of the investigator, might place the subject at unacceptable risk for participation in this study;
* Subjects with a history of cancer within the last five years (other than non-melanoma skin cell cancers cured by local resection). Existing non-melanoma skin cell cancers must be removed prior to dosing. Subjects with carcinoma in situ, treated with definitive surgical intervention, are allowed;
* Subjects who have a history of drug or alcohol abuse;
* Subjects with any serious bacterial infection within the last 3 months (such as pneumonia or pyelonephritis, unless treated and resolved with antibiotics);
* Subjects with serious, chronic or recurrent bacterial infection (such as recurrent pneumonia and chronic bronchiectasis);
* Subjects at risk for tuberculosis (TB), Specially, :

  1. Having evidences of clinical, imaging or lab test of current active or latent pulmonary tuberculosis;
  2. Having active pulmonary tuberculosis during the past 3 years, even if had treated;
  3. Having history of active pulmonary tuberculosis more than 3 years ago, unless the appropriate duration and types of anti-tuberculosis drug is well documented;
* Subjects with herpes zoster that resolved less than 2 months before enrollment;
* Subjects with evidence (as assessed by the Investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of Human Immunodeficiency Virus (HIV) infection;
* Subjects are impaired, incapacitated, or incapable of completing study related assessment;
* Hepatitis-B surface antigen-positive subjects.
* Hepatitis C antibody-positive subjects
* HIV antibody-positive subjects
* Subjects with any of the following laboratory values:

  1. Hgb < 85 g/L
  2. white blood cell count < 3,000/mm3(3×10^9/L)
  3. Platelets < 100,000/mm3(100×10^9/L);
  4. Creatinine clearance < 40 mL/min;
  5. Serum glutamic pyruvic transaminase (GPT or ALT) or glutamic oxaloacetic transaminase (GOT or AST)>2 times upper limit of normal;
  6. Any other laboratory test results that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in this study;
* Subjects who have received treatment with rituximab at any time;
* Subjects who had prior exposure to abatacept or CTLA4-Ig;
* Subjects who have received treatment with any investigational drug within 28 days (or less than 5 terminal half-lives of elimination) (whichever is longer);
* Subjects currently (when signing informed consent) treated with an anti-tumor necrosis factor (TNF) therapy, such as adalimumab and infliximab (within 8 weeks of the last dose), or etanercept (within 4 weeks of the last dose);
* Subjects who discontinued an approved biologic RA therapy due to lack of efficacy in the past;
* Subjects exposed to multiple (>3) approved biologic RA therapies in the past;
* Subjects currently treated with anakinra unless a minimum 4-week wash-out period has been completed before Day 1;
* Subjects who received prior treatment with any investigational biologic not currently approved;
* Subjects who had been exposed to any approved biologic within 4 weeks or 5 half-lives, whichever was longer;
* Subjects are (when signing informed consent)receiving an investigational biologic RA therapy or an approved biologic RA therapy;
* Subjects who have received any active vaccine within 3 months of the first dose of the study medication or plan to receive active vaccine during the study;
* Prisoners or subjects who are involuntarily incarcerated;
* Subjects who are compulsorily detained for treatment either a psychiatric or physical (e.g., infectious disease) illness;
* Subjects who are illiterate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects meeting ACR 20 at 24 weeks (Day 169) | Day 169
  The ACR 20 definition of improvement is a 20% improvement from baseline in the number of tender and swollen joints, and a 20% improvement from baseline in 3 of the remaining 5 core set measures: participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function and acute phase reactant value (C-reactive protein).

SECONDARY OUTCOMES:
The proportion of subject meeting Health Assessment Questionnaire Disability Index (HAQ-DI) improvement at 24 weeks (Day 169) | Day 169
  The HAQ questionnaire includes 20 questions to assess physical function in 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and common activities. The domain questions are evaluated on a 4-point scale: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty, 3=unable to do. A disability index was calculated by summing the worst scores in each domain and dividing by the number of domains answered. Clinically meaningful HAQ-DI response=an improvement of at least 0.3 units from baseline in HAQ-DI.
The proportion of subjects meeting ACR 50 at 24 weeks (Day 169) | Day 169
  The ACR 50 definition of improvement is a 50% improvement from baseline in the number of tender and swollen joint counts, and a 50% improvement from baseline in 3 of the remaining 5 core set measures: participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function and acute phase reactant value (C-reactive protein).
The proportion of subjects meeting ACR 70 at 24 weeks (Day 169) | Day 169
  The ACR 70 definition of improvement is a 70% improvement from baseline in the number of tender and swollen joint counts, and a 70% improvement from baseline in 3 of the remaining 5 core set measures: participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function and acute phase reactant value (C-reactive protein).

OTHER OUTCOMES:
The mean change of disease activity score from baseline by measuring DAS28-CRP at 24 weeks (Day 169) | Day 169
  The DAS28 index measures disease activity in rheumatoid arthritis and is a composite derived from the number of swollen/tender joints, laboratory tests of inflammation (C-reactive protein measured in mg/L), and participant assessment of global health (by marking a visual analog scale 100 mm line from "very good" to "very bad"). A higher DAS28 score indicates worse control of disease. High disease activity is > 5.1, low disease activity is < 3.2 and remission is < 2.6.
The mean change of HAQ-DI from baseline at 24 weeks (Day 169) | Day 169
Cmin of abatacept 125 mg administered SC weekly | Day1 to Day196 in double-blind period
Cmax of abatacept 125 mg administered SC weekly | Day71 to Day78 in open-label period
Area Under Curve (AUC) of abatacept 125 mg administered SC weekly | Day71 to Day78 in open-label period
Anti-abatacept antibodies | Day1 to Day421
Anti cytotoxic T lymphocyte-associated antigen-4(CTLA-4) antibodies | Day1 to Day421

CONTACTS AND LOCATIONS:
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No